CLINICAL TRIAL: NCT01576445
Title: Randomised Controlled Trial to Compare the Speed of Recovery and Functional Outcome Following Total Knee Replacement (TKR) Using a Quadriceps Sparing Approach to the Knee Against a Standard Medial Parapatellar Surgical Exposure
Brief Title: Functional Outcome in Two Types of Total Knee Replacement Surgery for People With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: DePuy International (Industry); Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Marietta van der Linden, Research Fellow Physiotherapy, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIS1
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; function
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mid-vastus approach (Experimental)
  Interventions: Procedure: Mid-vastus approach
- medial parapatellar approach (Experimental)
  Interventions: Procedure: medial parapatellar approach

INTERVENTIONS:
Procedure: Mid-vastus approach — Mid-vastus approach to avoid patellar eversion and to minimise the muscle split.
  Arms: Mid-vastus approach
Procedure: medial parapatellar approach — medial parapatellar approach
  Arms: medial parapatellar approach

SUMMARY:
When performing total knee replacement surgery, the surgeon has a choice as to which type of surgical technique to use. The standard technique at the Royal Infirmary in Edinburgh is the so-called 'medial parapatellar' exposure. And alternative and more recently introduced technique is the 'Mid-vastus approach' in which the surgeon will cut through less of the muscle at the front of the leg. In this study we compare the two surgical techniques in a so-called randomized trial. This means that we put people randomly into two groups, one group will receive surgery with the 'Mid-vastus approach' and the other group the surgery with the 'Medial parapatellar approach'. It is hypothesized that people who receive the Mid-vastus approach recover quicker and have a better short-term functional outcome than people who receive the 'Medial parapatellar approach'.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled double blind trial in which both immediate post-operative recovery and functional outcome at 6 weeks, 3 and 6 months after total knee replacement surgery will be assessed for two different types of surgical approach; Medial Parapatellar and Mid-vastus.

Functional outcome will be assessed by recording the kinematics of the lower limb joints in addition to muscle activity (electromyography) during walking, stair ascending and descending and getting up from a chair through computerized 3D motion analysis. Outcome measures will be recorded immediate post surgery and at medium follow-up and will cover all areas of the World Health Organisation, International Components of Functioning, Disability and Health (ICF) components 'Body Structures and Functions/Impairments' ,'Activities and Participation' and 'Personal factors'. It is hypothesized that by minimizing the damage to the quadriceps, patients operated using the Mid-vastus approach will have better muscle function and will therefore have more normal knee range of motion, knee joint loading and muscle activity patterns compared to those with the Medial Parapatellar approach.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty
* Osteoarthritis
* Surgery at Royal Infirmary Edinburgh by participating surgeons

Exclusion Criteria:

* A Body Mass Index of more than 40
* Fixed valgus deformity of more than 15 degrees
* Inflammatory polyarthritis
* disorders of the feet, ankles or hips or spine causing abnormal gait or significant pain
* dementia
* severe visual impairment
* neurological conditions affecting movement
* inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change in Functional knee range of motion from pre surgery to 6 months post surgery | 6 months after surgery
  The knee range of motion during functional activities such as walking and stair ascending and descending is recorded using three dimensional motion analysis

SECONDARY OUTCOMES:
change in WOMAC from pre surgery to 6 month after surgery | 6 months after surgery
  Western Ontario McMaster Universities (WOMAC) osteoarthris Index is patient-reported outcome and has three components: Pain, Stiffness and Function.
Change in Timed up and Go test from pre-surgery to 6 month post surgery | 6 months after surgery
Change in range of motion of the knee in prone from pre surgery to post surgery | 6 months after surgery
  The range of motion of the knee is measured using a manual goniometer.
Change in Objective daily physical activity from pre to 6 month post surgery | 6 month post surgery
  Objective daily physical activity is recorded using an activity monitor
Change in knee extensor strength from pre surgery to 6 months after surgery | 6 months after surgery
  Knee extensor strength is measured using a digital myometer

CONTACTS AND LOCATIONS:
Locations (1):
- New Royal infirmary Edinburgh, Edinburgh, United Kingdom